CLINICAL TRIAL: NCT03195816
Title: Effects of a Computer-based Cognitive Stimulation on the Verbal Learning and the Progression of White Matter Hyperintensities in Mild Cognitive Impairment: A Protocol for a Randomized Controlled Trial.
Brief Title: A Computer-based Cognitive Stimulation in Mild Cognitive Impairment With White Matter Hyperintensities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leila DJABELKHIR (Other)
Responsible Party: Sponsor-Investigator, Leila DJABELKHIR, PhD candidate, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUS3WMH
Record Dates: First submitted 2017-06-14; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; white matter hyperintensities; computerized cognitive training; brain plasticity
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Comparison between experimental group and control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computerized Cognitive training (Experimental): Experimental group will receive 1 year of a computer-based cognitive stimulation program.
  Interventions: Behavioral: Computerized Cognitive training
- MCI control group (No Intervention): The control group will receive a usual standard care without engagement in intervention

INTERVENTIONS:
Behavioral: Computerized Cognitive training — Experimental group will receive 1 year of a computer-based cognitive stimulation program, first 6 months, 60-minutes twice a week and next 6 months once a week training in group-setting, using a tablet with a software with specific training focused on attention, executive and speed processing functions.
  Arms: computerized Cognitive training

SUMMARY:
This is a non-pharmacological study evaluating the impact of a computerized cognitive stimulation program on verbal learning and on the progression white matter hyperintensities in elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
White matter hyperintensities (WMH) can appear in Mild Cognitive Impairment (MCI) and have been associated to executive, attention and processing speed deficits. Some findings indicate that the presence of WMH may contribute to Alzheimer's disease (AD) in addition to ß-amyloid, suggesting a greater vulnerability of MCI. One important challenge is to prevent or slowing down the progression of WMH. Few studies investigated the effects of computerized cognitive interventions in MCI with WMH, which deserve special attention. This study aim to investigate the effects of an intensive computer-based cognitive stimulation (CCS) program on the verbal learning in episodic memory in MCI with WMH and to explore the effects on the progression of WMH at 1-year interval.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* With and without with matter hyperintensities
* MRI data available or accept to perform one
* No engagement in other cognitive intervention program

Exclusion Criteria:

* Psychiatric and neurological disorders
* History of alcohol or other substance consumption
* Sensory and or motor deficit that could interfere with the use of computer tool
* Refusal MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change on Rey Auditory Verbal Learning test | Baseline assessment in 3-weeks period before intervention, change from baseline at 6-months immediately after the end intervention, and after 3-months follow-up
  Assessment of verbal learning in episodic memory

SECONDARY OUTCOMES:
Change on Fazekas scale | Baseline assessment of WMH severity and evolution at 12 months immediately after intervention
  Assessment of white matter hyperintentisites severity on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie AR RIGAUD, Professor, Principal Investigator — Broca University Hospital

IPD SHARING:
Plan to Share IPD: No